CLINICAL TRIAL: NCT03985800
Title: Specialty Medical Homes to Improve Outcomes for Patients With IBD and Behavioral Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mount Sinai Hospital, New York (Other); The Cleveland Clinic (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Eva Szigethy, Professor of Psychiatry and Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19020176; IHS-2017C3-8930 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2019-05-28; First posted 2019-06-14 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease; Behavioral Symptoms
MeSH Terms: conditions — Inflammatory Bowel Diseases; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: Comparison between technology interventions and in-person interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAM-care as usual approach (Active Comparator): Patients will be triaged based on their physical health (PH) and behavioral health (BH) complexity to determine the frequency of in-person visits and how much of these visits will be devoted to medical versus BH issues. Minor modifications were made to the TEAM approach during the COVID-19 public health emergency to account for reduced face-to-face time without changing the underlying differentiation between the two models of delivering SMH care.
  Interventions: Other: TEAM
- TECH-telehealth approach (Active Comparator): Each patient will have an initial face-to-face visit with the core treatment team described above and undergo the same triage process to determine their PH/BH care needs. Each TECH patient will participate in one face-to-face treatment team visit per year unless more frequent visits are deemed to be medically necessary; however, all other interactions will be conducted via technology-supported modalities
  Interventions: Other: TECH

INTERVENTIONS:
Other: TEAM — TEAM incorporates team-based care with traditional in-person clinic visits. The care team includes a gastroenterologist, nurse practitioner, nutritionist, social worker/behavioral health specialist, and a psychologist or psychiatrist.
  Arms: TEAM-care as usual approach
Other: TECH — TECH uses team-based care similar to TEAM, but in-person care is substituted with telemedicine (i.e., video visits and consultations) and digital behavioral health tools.
  Arms: TECH-telehealth approach

SUMMARY:
A comparative effectiveness study using an individual-level randomized design along with a pragmatic, mixed-methods approach to compare two strategies (e.g. in-person supported care, technology-supported care) all of which include evidence-based components for delivering IBD and BH care. Quantitative (e.g. self-report, electronic health record, process) and qualitative (e.g., interviews) data will be collected across multiple time points during the study period.

DETAILED DESCRIPTION:
The investigators propose to conduct a comparative effectiveness research (CER) study of two evidence-based, patient-centered approaches implemented within an existing Specialty Medical Home (SMH) model: TEAM, an in-person, multidisciplinary team-based approach delivered at point of care and TECH, a technology-based (digital therapeutics, and telehealth) approach delivered at the patient's convenience with the guidance of health coaches. Both are designed to support care for adult patients with complex, chronic health conditions and behavioral health (BH) disorders, and will be tested in three of the nation's largest and most established SMHs for inflammatory bowel disease (IBD). IBD serves as an exemplary chronic disease model where untreated BH issues have been associated with poor medical outcomes.

Primary outcomes are composite scores of measures focused on 1) IBD Symptom Severity, and 2) BH Symptom Severity. IBD Symptom Severity is measured via a composite IBD Complexity Score involving responses to two patient-reported scales: the PROMIS-GI measure and either the Harvey Bradshaw Index (for participants with Crohn's disease) or ulcerative colitis activity index (for participants with ulcerative colitis). BH Symptom Severity was measured utilizing the Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS), a composite of two patient-reported scale for measuring anxiety (Generalized Anxiety Disorder scale (GAD-7) and depression (Patient Health Questionnaire depression scale (PHQ-8). Scales are further defined in Results, Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel Disease Diagnosis of Crohn's or Ulcerative Colitis. Behavioral health symptoms mild to severe, defined as a score of >= 6 on the Personal Health Questionnaire 4 (PHQ4)

Exclusion Criteria:

* Lack of smart phone, and/or are unable to speak, read or understand English at the minimum-required level.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 657 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared. Data is shared at the aggregate level

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on July 1, 2019 and was completed on February 28, 2024. A brief pause in recruitment occurred between March 13 and September 13, 2020 to account for disruptions related to the COVID-19 pandemic. All participants were recruited from one of three specialty medical home clinics at large urban academic centers in the northeastern US: UPMC in Pittsburgh, Mount Sinai Hospital in New York, and the Cleveland Clinic in Cleveland.
Pre-assignment Details: All participants were randomly assigned to one of the two intervention arms upon successful enrollment in the study. Allocation was stratified based on age (18-30 or 31-60), IBD diagnosis (Crohn's disease or ulcerative colitis) and disease activity (low or high).
Groups:
- TEAM: TEAM is a high-human touch, multidisciplinary specialty medical home approach that connects participants with a personalized care team including gastroenterologists, advanced practice providers, behavioral health specialists, dietitians, registered nurses, pharmacists, and health coordinators who provide intensive support and resources for patients.
- TECH: TECH is a low-human touch approach leveraging behavioral digital tools - primarily a digital cognitive behavioral therapy mobile application with embedded health coaches - to deliver behavioral health care at the patient's convenience.
Period: Overall Study
Arm/Group | TEAM | TECH
Started | 329 | 328
Completed | 323 | 320
Not Completed | 6 | 8
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in baseline analysis.
Groups:
- TECH: TECH is a low-human touch approach leveraging behavioral digital tools - primarily RxWell, a digital cognitive behavioral therapy mobile application with embedded health coaches - to deliver behavioral health care at the patient's convenience.
- Total: Total of all reporting groups
Arm/Group | TEAM | TECH | Total
Number analyzed (Participants) | 329 | 328 | 657
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/gender self-reported by participants at baseline.
  Participants
    Gender: Female | 211 | 213 | 424
    Gender: Male | 93 | 90 | 183
    Gender: Other | 2 | 1 | 3
    Gender: Prefer not to answer | 1 | 1 | 2
    Gender: Missing | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity self-reported by participants at baseline.
  Participants
    Hispanic or Latino | 17 | 13 | 30
    Not Hispanic or Latino | 269 | 275 | 544
    Unknown or Not Reported | 43 | 40 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race self-reported by participants at baseline.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 6 | 3 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 24 | 13 | 37
    White | 254 | 271 | 525
    More than one race | 5 | 11 | 16
    Unknown or Not Reported | 40 | 30 | 70
IBD Diagnosis [Count of Participants; unit: Participants] — IBD diagnosis confirmed by physician at baseline.
  Participants
    Crohn's disease | 222 | 218 | 440
    Ulcerative colitis | 107 | 110 | 217
Steroid Use [Count of Participants; unit: Participants] — Incidence of steroid prescription at baseline was extracted from the electronic medical record.
  Participants
    Yes | 121 | 119 | 240
    No | 208 | 209 | 417
Opioid use [Count of Participants; unit: Participants] — Incidence of opioid prescription at baseline was extracted from the electronic medical record.
  Participants
    Yes | 108 | 105 | 213
    No | 216 | 218 | 434
    Missing | 5 | 5 | 10
Advanced therapy [Count of Participants; unit: Participants] — Incidence of advanced IBD therapy prescription at baseline was extracted from the electronic medical record. Advanced therapies include: Infliximab/Remicade, Adalimumab/Humira, Certolizumab/Cimzia, Golimumab/Simponi, Vedolizumab/Entyvio, Natalizumab/Tysabri, Ustekinumab/Stelara, Tofacitinib/Xeljanz, and Ozanimod/Zyposia.
  Participants
    Yes | 185 | 169 | 354
    No | 144 | 159 | 303
Comorbidity [Count of Participants; unit: Participants] — Incidence of any one of 14 investigator-defined select comorbidities at baseline. Comorbidities of interest include: AIDS; autonomic disorder; chronic kidney disease; chronic pain syndrome; connective tissue disease; COVID-19; diabetes (Type 1 or 2); irritable bowel syndrome; liver disease; peptic ulcer disease; primary sclerosing cholangitis; rheumatologic disease; short gut syndrome; and systemic autoimmune conditions.
  Participants
    Yes | 147 | 143 | 290
    No | 182 | 185 | 367
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of participants at baseline.
  Years | 34.7 (10.6) | 34.9 (10.8) | 34.8 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: IBD Symptom Severity
Description: IBD symptom severity was measured via a composite IBD Complexity Score developed by clinical researchers to quantify both biological and psychosocial domains of IBD within an SMH setting. It includes the sum of patient-reported responses to two scales: the PROMIS GI symptoms scale, evaluating four domains of gastrointestinal symptoms; and disease-specific PRO-2 disease severity indices taken from the Harvey Bradshaw Index (for individuals with Crohn's disease) and Ulcerative Colitis Activity Index (for individuals with ulcerative colitis). The complexity score is calculated by adding the value of the patient's PRO-2 to the cumulative PROMIS-GI score. Lower scores indicate lower symptom severity; higher scores indicate higher symptom severity. The minimum score is 0; the maximum score is open-ended based on patient response. Only the total IBD Complexity Score is reported.
Time Frame: Compare scores at Baseline, 6-month and 12-month for any changes
Population: Participants were included in the analysis for IBD Symptom Severity as long as they had complete covariate data and the IBD Complexity Score measured at at least one timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 75.9 (31.0) | 79.9 (31.3)
  Score at 6-month follow-up | 63.5 (30.0) | 65.0 (33.2)
  Score at 12-month follow-up | 62.3 (31.2) | 64.4 (32.2)
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of IBD complexity score does not differ by treatment group; Test type: Superiority — We calculated statistical power for the target sample size of 675 (~337 in each of TEAM and TECH arms). After adjusting for the multiple testing in Aim 1 (2 tests) and considering 25% attrition, a sample size of 505 (~252 per treatment group) will provide over 99.9% power for the hypothesis test for Aim 1; p = 0.53, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 1.26 with two degrees of freedom; Type III Wald chi-squared = 1.26
Statistical Analysis 2: Comparison: TEAM vs TECH; Aim 2b., moderation by age. Null hypothesis: Age does not moderate the trajectory of complexity score by treatment group; Test type: Superiority — Considering a range of effect sizes for B1, B2, and B3, we estimated the outcome Y as Y=B1*X+B2*M+B3*X*M+ε, where ε~N(0,1). Using Monte Carlo methods, we averaged across scenarios to determine the typical effect of B3 that can be detected with our current and projected sample sizes after 25% attrition. With our projected sample sizes we expect 0.80 power to detect a significant interaction when the magnitude of B3 is at least 0.50; p = 0.57, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time*age interaction term is 1.14 with two degrees of freedom; Type III Wald chi-squared = 1.14
Statistical Analysis 3: Comparison: TEAM vs TECH; Aim 2b., moderation by diagnosis. Null hypothesis: Diagnosis does not moderate the trajectory of complexity score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.96, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time*diagnosis interaction term is 0.08 with two degrees of freedom; Type III Wald chi-squared = 0.08
Statistical Analysis 4: Comparison: TEAM vs TECH; Aim 2b., moderation by site. Null hypothesis: Site does not moderate the trajectory of complexity score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.17, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time*site interaction term is 6.41 with two degrees of freedom; Type III Wald chi-squared = 6.41
Statistical Analysis 5: Comparison: TEAM vs TECH; Aim 2b., moderation by eHealth literacy. Null hypothesis: eHealth literacy does not moderate the trajectory of complexity score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.27, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time*site interaction term is 2.6 with two degrees of freedom; Type III Wald chi-squared = 2.6

2. Primary Outcome: Behavioral Health Symptom Severity
Description: Behavioral health symptom severity was measured utilizing the Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) - which combines the PHQ-8 and GAD-7 scales - as a composite measure of depression and anxiety. The Patient Health Questionnaire 8-item depression scale (PHQ-8) and 7-item Generalized Anxiety Disorder scale (GAD-7) are among the best validated and most commonly used depression and anxiety measures, respectively. The PHQ-ADS is the sum of the PHQ-8 and GAD-7, where a decrease in scores indicates a decrease in BH symptom severity; a decrease of 3-4 points indicates MCID. Lower scores indicate lower levels of behavioral health symptom severity; higher scores indicate higher symptom severity. The minimum score is 0; the maximum score is 45. Only the total PHQ-ADS is reported.
Time Frame: Compare at Baseline, 6-month and 12-month for any changes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 25.4 (7.88) | 26.2 (7.94)
  Score at 6-month follow-up | 18.7 (10.9) | 19.7 (10.9)
  Score at 12-month follow-up | 18.0 (11.2) | 19.2 (11.5)
Statistical Analysis 1: Comparison: TEAM vs TECH; Aim 1. The trajectory of PHQ-ADS does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.90, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 0.21 with two degrees of freedom; Type III Wald chi-squared = 0.21
Statistical Analysis 2: Comparison: TEAM vs TECH; Aim 2a, moderation by disease activity. Null hypothesis: Disease activity does not moderate the trajectory of behavioral health score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.55, Mixed Models Analysis — Threshold for statistical significance was 0.05; Type III Wald chi-squared = 1.21
Statistical Analysis 3: Comparison: TEAM vs TECH; Aim 2b, moderation by age. Null hypothesis: Age does not moderate the trajectory of behavioral health score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.50, Mixed Models Analysis — Threshold for statistical significance was 0.05; The Chi-squared statistic for the group*time*age interaction term is 1.37 with two degrees of freedom; Type III Wald chi-squared = 1.37
Statistical Analysis 4: Comparison: TEAM vs TECH; Aim 2b, moderation by diagnosis. Null hypothesis: Diagnosis does not moderate the trajectory of behavioral health score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.08, Mixed Models Analysis — Threshold for statistical significance was 0.05; The Chi-squared statistic for the group*time*diagnosis interaction term is 5.16 with two degrees of freedom; Type III Wald chi-squared = 5.16
Statistical Analysis 5: Comparison: TEAM vs TECH; Aim 2b, moderation by site. Null hypothesis: Site does not moderate the trajectory of behavioral health score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 1.0, Mixed Models Analysis — Threshold for statistical significance was 0.05; The Chi-squared statistic for the group*time*site interaction term is 0.11 with two degrees of freedom; Type III Wald chi-squared = 0.11
Statistical Analysis 6: Comparison: TEAM vs TECH; Aim 2b, moderation by eHealth literacy. Null hypothesis: eHealth literacy does not moderate the trajectory of behavioral health score by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.20, Mixed Models Analysis — Threshold for statistical significance was 0.05; The Chi-squared statistic for the group*time*eHealth literacy interaction term is 3.23 with two degrees of freedom; Type III Wald chi-squared = 3.23

3. Secondary Outcome: Functional Impairment
Description: Functional impairment was measured using the validated Short Form 12 Health Survey Version 2 (SF-12v2) which includes 12 items from the Short-Form 36 Health Survey and yields a physical and mental composite score as well as 8 subscale values: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Responses are tallied via a norm-based scoring algorithm provided by the assessment licensing company. Lower scores correspond with poorer health-related functioning; higher scores indicate better health-related functioning. The minimum score is 18.5; the maximum score is 142.6. Only the total composite score (the sum of both the physical and mental scales) is reported.
Time Frame: Compare at baseline, 6-month and 12-month for any changes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 37.6 (6.57) | 38.4 (6.36)
  Score at 6-month follow-up | 34.2 (7.98) | 34.7 (7.58)
  Score at 12-month follow-up | 33.3 (7.70) | 33.5 (8.07)
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of functional impairment does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.53, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 3.09 with two degrees of freedom; Type III Wald chi-squared = 3.09

4. Secondary Outcome: IBD-IBS Symptom Severity
Description: IBD-IBS Symptom Severity was measured using the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) to more accurately capture IBD symptom severity for many individuals with IBD, particularly those with inactive IBD but persistent functional GI symptoms (e.g., IBD-IBS). The IBS-SSS scores pain severity, pain frequency, abdominal bloating, bowel satisfaction and interference with life on a 0-100 scale with a total score of 500. A 50-point or more reduction in this score is considered clinically meaningful. Total scores range from 0 to 500 with higher scores indicating more severe symptoms. Answers to all questions are summed to achieve the total score. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS. Only total scores are reported.
Time Frame: Compare at baseline, 6-month and 12-month for any changes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 222 (135) | 238 (130)
  Score at 6-month follow-up | 185 (125) | 175 (123)
  Score at 12-month follow-up | 174 (124) | 179 (125)
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of IBD-IBS symptom severity does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 6.01 with two degrees of freedom; Type III Wald chi-squared = 6.01

5. Secondary Outcome: Health Care Utilization
Description: Health care utilization was captured through EHR data to measure categorical (yes or no) instances of ED visits and inpatient hospitalizations at both 6- and 12-months post-enrollment.
Time Frame: Compare at baseline, 6-month and 12-months for any changes
Measure: Count of Participants; unit: Participants
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Participants
  Hospitalizations: Yes | 35 | 36
  Hospitalizations: No | 292 | 291
  Hospitalizations: Missing | 2 | 1
  ED Visits: Yes | 27 | 31
  ED Visits: No | 297 | 297
  ED Visits: Missing | 5 | 0
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of hospitalizations does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.13, Mixed Models Analysis — The threshold for statistical significance was .05; For hospitalizations, the Chi-squared statistic for the group*time interaction term is 4.14 with two degrees of freedom; Type III Wald chi-squared = 4.14
Statistical Analysis 2: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of ED visits does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.67, Mixed Models Analysis — The threshold for statistical significance was .05; For ED visits, the Chi-squared statistic for the group*time interaction term is 0.82 with two degrees of freedom; Type III Wald chi-squared = 0.82

6. Secondary Outcome: Patient Engagement
Description: Patient engagement was measured using the validated IBD Self-Efficacy Scale (IBD-SES) which assesses one's confidence level in managing stress and emotions, managing medical care, managing symptoms and disease, and maintaining remission. The IBD-SES measures self-management activities across four subscales (Stress and Emotions; Medical Care; Symptoms and Disease; Remission), with higher scores indicating greater confidence in self-management. Responses for each question are summed to produce one overall and four subscale scores. The total score range is between 29 and 290, with 29 indicating the lowest level of self-efficacy and 290 indicating the highest. Each item is scored 1-10, with 1 being assigned for responses of "Not confident at all" and a score of 10 assigned for responses of "Totally confident." Only total scores are reported.
Time Frame: Compare at baseline, 6-month and 12-month for any changes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 161 (40) | 157 (35.8)
  Score at 6-month follow-up | 174 (47.5) | 178 (46.9)
  Score at 12-month follow-up | 178 (54.0) | 178 (49.7)
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of self-efficacy does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.37, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 1.98 with two degrees of freedom; Type III Wald chi-squared = 1.98

7. Secondary Outcome: Quality of Life
Description: Quality of life was evaluated using the Short Quality of Life in Inflammatory Bowel Disease Questionnaire (SIBDQ), a validated tool which measures physical, social, and emotional health-related quality of life (QOL) for patients with Crohn's disease and ulcerative colitis. On a 7-point scale, lower scores correspond with a lower perceived QOL, while higher scores represent a higher perceived QOL. Responses for each question are summed for a total score between 10 and 70, with 10 reflecting poor QOL and 70 reflecting high QOL. Each item is scored 1-7, with 1 being assigned for responses indicating the highest severity of symptoms, and 7 being assigned for those reflecting the lowest severity of symptoms. Only total scores are reported.
Time Frame: Compare at baseline, 6-month and 12-month for any changes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TEAM | TECH
Number analyzed (Participants) | 329 | 328
Score on a scale
  Score at baseline | 37.7 (10.7) | 35.5 (10.7)
  Score at 6-month follow-up | 42.6 (12.0) | 41.4 (11.9)
  Score at 12-month follow-up | 43.0 (12.5) | 43.4 (12.4)
Statistical Analysis 1: Comparison: TEAM vs TECH; Null hypothesis: The trajectory of quality of life does not differ by treatment group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.06, Mixed Models Analysis — The threshold for statistical significance was .05; The Chi-squared statistic for the group*time interaction term is 5.57 with two degrees of freedom; Type III Wald chi-squared = 5.57

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up (12 months after enrollment)
Description: All enrolled participants were included in the analysis population for adverse events. Adverse events align with ClinicalTrials.gov definitions.
Arm/Group | TEAM | TECH
All-Cause Mortality (participants affected / at risk) | 1/329 | 2/328
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/328
Other Adverse Events (participants affected / at risk) | 0/329 | 0/328

LIMITATIONS AND CAVEATS:
Sensitivity analyses confirmed that the COVID-19 pandemic did not have a significant impact on outcomes. Heterogeneity of patient and clinical factors could have introduced confounders that were not the focus of our primary analyses (e.g. specific comorbid medical diagnoses, the contribution of pharmacological treatment). Adherence/dose-effect was not examined beyond exploratory per-protocol analyses. Longer-term follow-up may have been needed to show impact on healthcare utilization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03985800/Prot_SAP_000.pdf